CLINICAL TRIAL: NCT00718510
Title: A Randomised, Double-blind, Cross-over, Placebo Controlled, Adjunctive-treatment of L-arginine Added to Treatment-as-usual (TAU) in Schizophrenia
Brief Title: L-arginine in Treatment as Usual in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Serdar Dursun, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPAT7176
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-arginine first/placebo second (Active Comparator): Patients with diagnosis of schizophrenia will be randomised to receive L-arginine first/placebo second 3 grams bid (cross-over design) in addition to treatment as usual. The active treatment period will be 3 weeks, with a wash-out period of 5 days and re-commencing on the alternative arm of the randomization
  Interventions: Drug: L-Arginine
- Placebo first/L-arginine second (Placebo Comparator): Patients with diagnosis of schizophrenia will be randomised to receive placebo first/L-arginine second 3 grams bid (cross-over design) in addition to treatment as usual. The active treatment period will be 3 weeks, with a wash-out period of 5 days and re-commencing on the alternative arm of the randomization
  Interventions: Drug: L-Arginine

INTERVENTIONS:
Drug: L-Arginine — 3 grams, twice daily, oral administration
  Other Names: Placebo

SUMMARY:
STUDY OBJECTIVES: To determine whether the addition of L-arginine to treatment as usual (TAU) in schizophrenia further improves and enhances therapeutic efficacy (positive, negative and depressive symptoms) and effectiveness of antipsychotic treatment

STUDY POPULATION: Patients diagnosed (DSM-IV criteria) with schizophrenia or schizoaffective disorder

Total expected number of patients: 14

INVESTIGATIONAL COMPOUND: L-arginine capsules, 3 grams of L-arginine given twice a day (total daily dose of 6 grams/day)

DURATION OF ACTIVE TREATMENT: 3 weeks followed by wash-out phase of 5 days and 3 weeks of second treatment phase (cross-over design)

EVALUATION CRITERIA: Primary (efficacy) outcomes: PANSS scores. Secondary outcomes: Calgary Depression Scale for schizophrenia, CGI; AIMS, UKU-assessment of side-effects

ASSESSMENT SCHEDULE: Treatment arm 1: Baseline, weeks: 1,2,3, wash-out phase; week 4, cross-over phase: treatment phase-2; weeks 5,6,7

STATISTICAL CONSIDERATIONS: Analysis of variance of outcome measures with treatment as the between-subject factor and pre- and post-treatment scores as within- subjects factors.

DURATION OF STUDY PERIOD: Patient recruitment to be completed in 12 months, study full completion 18 months.

DETAILED DESCRIPTION:
In the current study, our goals were to examine the clinical benefits of the nitric oxide (NO) donor and main precursor of NO, L-arginine, to further improve the symptoms of schizophrenia with minimum or no additional side-effects. L-Arginine is classified as a semi-essential or conditionally essential amino acid depending on the developmental stage and health status of the individual. Glutamate N-methyl-D-aspartate (NMDA) receptors have functional connections to the NO system in the brain. Dysfunction of connectivity of the neuroregulators glutamate and NO have been implicated in mechanisms of psychosis. Therefore, any downstream effects of NMDA dysfunction in schizophrenia may be ultimately mediated by the NO system at a cellular level. As an augmenting treatment to antipsychotic therapy, we examined the ability of L-arginine to further improve residual symptoms in the illness.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Diagnoses of schizophrenia or schizoaffective disorder using the Diagnostic and Statistical Manual-IV (DSM-IV) criteria
3. Competent and willing to give informed consent
4. Able to take oral medication and likely to complete the required evaluations.
5. Medication remained stable 4 weeks prior to baseline.
6. Female participants of child bearing capability must be willing to use adequate contraceptives (4.6.1a) for the duration of the study, and, willing to have a pregnancy test pretreatment and during the study.

Adequate contraception is defined as use of contraceptive double barrier system (i.e. condom and spermicide) or contraceptive implant, oral contraceptive or injected depot contraceptive plus other form of contraceptive, i.e. condom. Females will be considered incapable of child bearing if they are one year postmenopausal or irreversibly surgically sterilised.

Exclusion Criteria:

* Relevant medical illness [serious renal, diabetes, hepatic, cardiac, low- or high-blood-pressure or other illnesses] in the opinion of the investigators. In particular, history of past or recent cardiac illness, MI and abnormal ECG and current treatments for cardiac illness. The results of the Laboratory Investigations (LFT, TFT, RFT, WBC, ECG, platelets, blood chemistry, lipids, weight/BMI) will be taken into account in determining the exclusion criteria.

  1. Relevant medical illness will be determined in the first instance by asking the patients mental health care team if the patient has any medical condition/problems. After consent has been obtained, the research nurse/research doctor will then have access to the patient's notes and if necessary communicate with his/her GP and will assess patient eligibility to take part in the clinical trial by scrutinising the patient's past medical history, most recent blood results, electrocardiograms, as well as any physical tests that have been performed on the patient. If there are any deviations from the 'norm' the investigators will assess the eligibility of the individual patient.
  2. Patients receiving active treatments for Herpes virus as L-arginine may counteract the benefits of lysine to treat herpes virus
  3. Patients who are currently receiving NSAIDs or other drugs that can cause significant stomach an gastrointestinal side-effects
  4. Drugs that alter potassium levels in the body, such as ACE inhibitors and potassium sparing diuretics
  5. Patients who are pregnant or plan to become pregnant while using this amino acid
  6. Patients who are breastfeeding
  7. Prior history of intolerance to L-arginine
  8. Any significant change of psychotropic medications done within the previous 4 weeks
  9. Diagnosis of substance abuse (except nicotine or caffeine) or dependence within the last three months according to DSM-IV criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Dursun, M.D., Ph.D., Principal Investigator — University of Alberta; Glen Baker, Ph.D., D.Sc., Principal Investigator — University of Alberta; John C. Lind, Ph.D., Principal Investigator — Alberta Hospital Edmonton; Phil Tibbo, F.R.C.P.C., Principal Investigator — University of Alberta; Mee-Sook Song, Ph.D., Principal Investigator — University of Alberta; Pierre Flor-Henry, F.R.C.P.C., Principal Investigator — Alberta Hospital Edmonton; Diane Cox, Ph.D., Principal Investigator — University of Alberta
Locations (1):
- Alberta Hospital Edmonton, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- L-arginine Treatment First, Placebo Treatment Second: The trial participants received 6 g p.o. (3 g twice per day at 0800h and 2000h) of L-arginine 500mg capsules for 3 weeks in addition to their antipsychotic treatment as usual. After a 5 day washout period, they then received placebo capsules (matching L-arginine 500mg) 6g p.o. (3 g twice per day at 0800h and 2000h) for 3 weeks in addition to their antipsychotic treatment as usual.
- Placebo Treatment First, L-arginine Treatment Second: The trial participants received the placebo capsules (matching L-arginine 500mg) 6 g p.o. (3 g twice per day at 0800h and 2000h) for 3 weeks in addition to their antipsychotic treatment as usual. After a 5 day washout period, they then received L-arginine (500mg capsules) 6g p.o. (3 g twice per day at 0800h and 2000h) for 3 weeks in addition to their antipsychotic treatment as usual.
Period: First Intervention (3 Weeks)
Arm/Group | L-arginine Treatment First, Placebo Treatment Second | Placebo Treatment First, L-arginine Treatment Second
Started | 7 | 8
Received Intervention (Received Intervention) | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (5 Days)
Arm/Group | L-arginine Treatment First, Placebo Treatment Second | Placebo Treatment First, L-arginine Treatment Second
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | L-arginine Treatment First, Placebo Treatment Second | Placebo Treatment First, L-arginine Treatment Second
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-arginine Treatment First, Placebo Treatment Second | Placebo Treatment First, L-arginine Treatment Second | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (15.1) | 37.8 (8.1) | 36 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Positive and Negative Syndrome Scale (PANSS) Total and Positive, Negative and General Psychopathology Subscale Scores at 3 Weeks
Description: The primary outcome measure was the Positive and Negative Syndrome Scale (PANSS) total score and PANSS positive, negative and general psychopathology subscale scores. The PANSS is a 30-item scale used to evaluate the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score (30 items) ranges from 30 to 210 with a higher score indicating a greater severity of symptoms. The PANSS positive symptom subscale score (7 items) ranges from 7=absent to 49=extreme; the PANSS negative subscale score (7 items) ranges from 7=absent to 49=extreme; and the PANSS general psychopathology subscare score (16 items) ranges from 16=absent to 112=extreme.
Time Frame: Baseline and 3 Weeks
Population: All participants who received all doses of each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- L-arginine: Participants who received L-arginine 6 g (500mg capsules) at 0800h and 2000h in either the first or last 3 weeks of the study
- Placebo: Participants who received Placebo 6 g (matching L-arginine 500mg capsules) at 0800h and 2000h in either the first or last 3 weeks of the study.
Arm/Group | L-arginine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  PANSS Total Score at Baseline | 71.6 (7.2) | 72.2 (5.7)
  PANSS Total Score at 3 Weeks | 68.0 (7.2) | 70.2 (7.0)
  PANSS Positive Scale at Baseline | 14.6 (4.4) | 14.3 (4.5)
  PANSS Positive Scale at 3 Weeks | 14.5 (4.6) | 13.6 (4.0)
  PANSS Negative Scale at Baseline | 22.8 (5.0) | 22.6 (4.3)
  PANSS Negative Scale at 3 Weeks | 21.9 (5.2) | 22.2 (5.2)
  PANSS General Psychopathology Score at Baseline | 33.4 (4.4) | 34.4 (2.7)
  PANSS General Psychopathology Score at 3 Weeks | 31.2 (3.9) | 33.6 (3.7)
Statistical Analysis 1: Comparison: L-arginine vs Placebo; Null hypothesis is that there was no difference in change of PANSS between L-arginine and Placebo. A two-factor ANOVA was used across all subjects with the within-subject factor being the treatment phase (L-arginine first/Placebo second or Placebo first/L-arginine second) and the between-subject factor being the day of treatment (time). A sample size of 14 patients was needed to give 90% power to detect a 4 point difference on the PANSS. This included a drop-out rate of about 10%; Test type: Other; p < 0.05, ANOVA — General Psychopathology Subscale Score; F(1,11)=5.03

2. Secondary Outcome: Change From Baseline in Mean Clinical Global Impression (CGI) Scale at 3 Weeks
Description: The Secondary Outcome Measure was the Clinical Global Impression (CGI) scale. The CGI is a 3-item scale that rates treatment response and monitors the clinical course of all psychiatric illnesses including schizophrenia. Within the CGI, the Severity of Illness was rated on a 7-point scale, 0=not assessed to 7=among the most severely ill patients. For Global Improvement, the total improvement following treatment as compared to at baseline of the trial was rated on a 7-point scale, 0=not assessed to 7=very much worse.
Time Frame: Baseline and 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-arginine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  CGI Score at Baseline | 4.0 (0) | 4.0 (0)
  CGI Score at 3 Weeks | 3.6 (0.5) | 3.7 (0.4)
Statistical Analysis 1: Comparison: L-arginine vs Placebo; Null hypothesis is that there was no difference in change of CGI ratings between L-arginine and Placebo. A two-factor ANOVA was used across all subjects with the within-subject factor being the treatment phase (L-arginine first/Placebo second or Placebo first/L-arginine second) and the between-subject factor being the day of treatment (time); Test type: Other; p = 0.46, ANOVA

3. Secondary Outcome: Change From Baseline in Mean Calgary Depression Scale for Schizophrenia (CDSS) at 3 Weeks
Description: The Secondary Outcome Measure was the Calgary Depression Scale for Schizophenia (CDSS). The CDSS is a 9-item scale that is used to rate the depressive symptoms in patients with schizophrenia. For each CDSS item, symptom severity was rated on a 3-point scale, from 0=absent to 3=severe. The CDSS total score ranges from 0 to 27 with a higher score indicating a greater severity of symptoms.
Time Frame: Baseline and 3 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-arginine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  CDSS at Baseline | 4.5 (3.4) | 4.5 (2.8)
  CDSS at 3 Weeks | 3.4 (2.7) | 3.8 (2.1)
Statistical Analysis 1: Comparison: L-arginine vs Placebo; Null hypothesis is that there was no difference in change of CDSS ratings between L-arginine and Placebo. A two-factor ANOVA was used across all subjects with the within-subject factor being the treatment phase (L-arginine first/Placebo second or Placebo first/L-arginine second) and the between-subject factor being the day of treatment (time); Test type: Other; p = 0.55, ANOVA

ADVERSE EVENTS:
Time Frame: Three weeks for each intervention
Description: Safety population included all participants that received at least one dose of the intervention
Arm/Group | L-arginine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No